CLINICAL TRIAL: NCT07342465
Title: Safety, Feasibility, and Preliminary Efficacy of Non-invasive Gamma Neuromodulation in Individuals With Schizophrenia Spectrum Disorders
Brief Title: Gamma Light and Sound Stimulation in Schizophrenia
Acronym: Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2505001650; Aging brain initiative (Other Grant/Funding Number: Massachusetts Institute of Technology)
Record Dates: First submitted 2025-11-21; First posted 2026-01-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia Spectrum Disorders
Keywords: schizophrenia; sensory stimulation; gamma stimulation; GENUS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Gamma Stimulation (Active Comparator): 40 Hz light and sound using GENUS device
  Interventions: Device: GENUS
- Sham Stimulation (Sham Comparator): Sham light and sound
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: GENUS — Sensory stimulation using light and sound
  Arms: Gamma Stimulation
Device: Sham Stimulation — Sham light and sound
  Arms: Sham Stimulation

SUMMARY:
Schizophrenia (SZ) is a severe neuropsychiatric disorder impacting over 20 million people globally, causing significant personal and societal burdens, particularly due to cognitive deficits and negative symptoms inadequately treated by current therapies. To address this gap, investigators propose using Gamma Entrainment Using Sensory Stimulation (GENUS), a novel, home-based treatment involving synchronized 40 Hz light-and-sound stimulation aimed at improving neural synchrony, cognition, and SZ symptoms. This innovative approach leverages advanced neurostimulation, biological, and neuroimaging methods to directly target gamma dysfunction, fulfilling an urgent need for effective and accessible at-home therapies.

The goal of this clinical trial is to learn about the safety and feasibility of gamma stimulation using light and sound. It will also learn if gamma stimulation using light and sound works to treat clinical symptoms and cognitive impairments in schizophrenia. The main questions it aims to answer are:

1. Is gamma stimulation safe for patients with schizophrenia spectrum disorders?
2. Does gamma stimulation alleviate clinical symptoms and cognitive impairments in schizophrenia patients?

Participants will:

1. Have an acute 1-hour stimulation at MIT.
2. Come for a one-day visit to MIT for stimulation, neuroimaging, clinical, and cognitive evaluations.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental illness that affects about half a percent of people worldwide. It can cause hallucinations, delusions, disorganized thoughts, reduced motivation, and problems with memory and concentration. While current medications can help with hallucinations and delusions, they are often less effective for improving thinking skills and motivation-two areas that strongly affect a person's daily life.

Scientists have found that people with schizophrenia often show changes in how their brain cells communicate and synchronize their activity. In particular, a type of brain rhythm called gamma oscillation-which normally helps with attention, memory, and perception-does not function properly. These rhythmic signals depend on a healthy balance between brain cells that excite and those that inhibit activity. When this balance is disrupted, it can lead to cognitive and emotional difficulties.

Our study focuses on a new non-invasive approach called Gamma Entrainment Using Sensory Stimulation (GENUS). GENUS uses light and sound flickering at 40 Hz (forty times per second) to gently stimulate the brain and restore its natural rhythmic patterns. Earlier studies have shown that this type of stimulation is safe, well-tolerated, and can improve brain activity and memory in people with Alzheimer's disease.

Because both Alzheimer's disease and schizophrenia involve similar problems with gamma rhythms, GENUS may also help improve brain function and symptoms in people with schizophrenia. This study will test whether 40 Hz light and sound stimulation is safe, feasible, and beneficial for individuals living with schizophrenia. Investigators aim to understand whether this type of sensory stimulation can enhance brain activity and support improvements in thinking and daily functioning

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-65 years of age.
2. A diagnosis of schizophrenia or schizoaffective disorder
3. No medication is an absolute exclusion. Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following: the patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS (central nervous system) active drugs.
4. The subject is willing to sign the informed consent document.
5. If the subject is deemed not to have the capacity to sign the informed consent, he/she will need a legally authorized representative to provide surrogate consent.

Exclusion Criteria:

1. Subjects who do not have healthcare
2. MRI contraindications such as the presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin or body.
3. High myopia < -7 diopters, or untreated cataracts that affect vision.
4. Clinical conditions:

   1. History of seizure or medical diagnosis of epilepsy.
   2. ECT history > 6 months
   3. Female subjects who are pregnant or currently breastfeeding.
   4. Longstanding premorbid history (i.e., longer than 10 years) of alcohol or substance abuse with continuous abuse up to and including the time that the symptoms leading to clinical presentation developed.
   5. Significant neurological or medical disorders that may produce cognitive impairment.
   6. Profound hearing or visual impairment.
   7. Eye surgery in the last 3 months or are scheduled to have eye surgery in the next 3 months (during the study)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety, feasibility, compliance | Immediately after the completion of stimulation
  Feasibility of gamma frequency stimulation in subjects with SZ will be assessed by analyzing the neurophysiological data from each subject for a sign of change in gamma frequency waves and determining the percentage of subjects who show this change.
  Tolerability and safety of gamma frequency stimulation will be assessed using questionnaires and measures to rate the subjects' overall experience with the stimulation. These questionnaires will monitor for any adverse effects of the stimulation.

SECONDARY OUTCOMES:
Changes in event related potentials and cognitive performance in 40 Hz ASSR, 2-back and Oddball tasks | Baseline and immediately after stimulation
Changes in neuroimgaing outcomes | Immediately after the completion of stimulation
  Changes in Glutamate and GABA using MRS and MRI

OTHER OUTCOMES:
Exploratory outcomes - Changes in the Positive and Negative Syndrome Scale | Immediately after the completion of stimulation
  Changes in the clinical symptoms assessment by the Positive and Negative Syndrome Scale
Exploratory outcomes - Changes in the Montreal Cognitive Assessment | Immediately after the completion of stimulation
  Changes in cognitive performance assessed by the Montreal Cognitive Assessment
Exploratory outcomes - Changes in Inflammatory markers | Immediately after the completion of stimulation
  Changes in Inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Li-Huei Tsai, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology (MIT), Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
All IPD collected throughout the trial, only IPD used in the results publication.

REFERENCES:
- [Result] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Result] Black T, Jenkins BW, Laprairie RB, Howland JG. Therapeutic potential of gamma entrainment using sensory stimulation for cognitive symptoms associated with schizophrenia. Neurosci Biobehav Rev. 2024 Jun;161:105681. doi: 10.1016/j.neubiorev.2024.105681. Epub 2024 Apr 17. PMID 38641090
- [Result] Chan D, Suk HJ, Jackson BL, Milman NP, Stark D, Klerman EB, Kitchener E, Fernandez Avalos VS, de Weck G, Banerjee A, Beach SD, Blanchard J, Stearns C, Boes AD, Uitermarkt B, Gander P, Howard M 3rd, Sternberg EJ, Nieto-Castanon A, Anteraper S, Whitfield-Gabrieli S, Brown EN, Boyden ES, Dickerson BC, Tsai LH. Gamma frequency sensory stimulation in mild probable Alzheimer's dementia patients: Results of feasibility and pilot studies. PLoS One. 2022 Dec 1;17(12):e0278412. doi: 10.1371/journal.pone.0278412. eCollection 2022. PMID 36454969